CLINICAL TRIAL: NCT01042093
Title: Efficacy of Multimodal Perioperative Analgesia Protocol With Periarticular Drug Injection in Total Knee Arthroplasty: A Randomized, Double Blind Study
Brief Title: Efficacy of Multimodal Perioperative Analgesia With Periarticular Drug Injection in Total Knee Arthroplasty(TKA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Towson Orthopaedic Associates (Other)
Responsible Party: Principal Investigator, David F. Dalury, MD, Orthopaedic Surgeon, Towson Orthopaedic Associates
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1113723
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Results first posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-09

CONDITIONS: Osteoarthritis,Knee
Keywords: Analgesia; postoperative pain; periarticular; arthroplasty; pain management
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia; Pain, Postoperative | interventions — Ropivacaine; Ketorolac Tromethamine; Clonidine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ROP/EPI/TOR/CLO (Active Comparator): Ropivacaine 5mg/ml (49.25 ml) Epinephrine 1 mg/ml (0.5 ml) Toradol 30mg/ml (1 ml) Clonidine 0.1 mg/ml (0.08mg - 0.8 ml)
  Interventions: Drug: Ropivacaine; Drug: Toradol; Drug: Clonidine; Drug: Epinephrine
- ROP/EPI/TOR (Active Comparator): Ropivacaine 5mg/ml (49.25 ml) Epinephrine 1 mg/ml (0.5 ml) Toradol 30mg/ml (1 ml)
  Interventions: Drug: Ropivacaine; Drug: Toradol; Drug: Epinephrine
- ROP/EPI/CLO (Active Comparator): Ropivacaine 5mg/ml (49.25 ml) Epinephrine 1 mg/ml (0.5 ml) Clonidine 0.1 mg/ml (0.08mg - 0.8 ml)
  Interventions: Drug: Ropivacaine; Drug: Clonidine; Drug: Epinephrine
- ROP/EPI (Active Comparator): Ropivacaine 5mg/ml (49.25ml) Epinephrine 1 mg/ml (0.5 ml)
  Interventions: Drug: Ropivacaine; Drug: Epinephrine

INTERVENTIONS:
Drug: Ropivacaine — Ropivacaine 5mg/ml (49.25 ml)
  Other Names: periarticular injection
Drug: Toradol — Toradol 30mg/ml (1 ml)
  Other Names: periarticular injection
  Arms: ROP/EPI/TOR; ROP/EPI/TOR/CLO
Drug: Clonidine — Clonidine 0.1 mg/ml (0.08mg - 0.8 ml)
  Other Names: periarticular injection
  Arms: ROP/EPI/CLO; ROP/EPI/TOR/CLO
Drug: Epinephrine — Epinephrine 1 mg/ml (0.5 ml)
  Other Names: periarticular injection

SUMMARY:
The purpose of this study is to compare different medication combinations used in a periarticular injection after total knee replacement surgery(TKR). A periarticular injection is an injection that is given into the tissues surrounding the knee joint. The injection is given while the patient is still in surgery.

The study will compare the level of pain management, length of hospital stay, range of motion and side effects from subjects receiving one of four different combinations of medication in a periarticular injection. The medications used in the injections are approved medications routinely used for pain management.

Approximately 160 subjects will participate in this study. The surgeon, study personnel, and patients will be blinded to the combination of medications each patient receives. The pharmacist will prepare the 4 different combinations of medications, randomize each patient to the particular combination of medications, and maintain the study drug documentation.

DETAILED DESCRIPTION:
Data Collection:

Data will be collected from the patient's pre-operative office visit, up to six weeks post-operatively.

Variables

Pre-operative Collection:

* Vital signs
* Hb/Hct
* Age
* Sex
* BMI
* WOMAC Score - Screen Failure at 36 or 12
* Visual Analog Scale (VAS)

Intra-operative Collection:

* Duration of surgery
* Tourniquet time
* Time of periarticular injection

Post-operative Collection:

* Pain Scores in the inpatient post-anesthesia care unit (PACU) using the 1- to 10- point Visual Analog Scale (VAS) an admission to unit, 1 hour, 2 hour, and on discharge.
* VAS pain scores every 8 hours on the Orthopaedic floor
* Use of supplementary narcotics
* Use of anti-emetics
* Serious Adverse Events (SAE) including deep vein thrombosis (DVT) formation, pulmonary embolism (PE), myocardial infarct or other serious cardiac event, excessive bleeding
* Length of hospital stay
* Requirement for inpatient rehabilitation versus discharge home
* Hours/Days to straight leg raise -POD 1, 2, 3 by MD on rounds.
* Days to independent ambulation
* Hemoglobin and Hematocrit levels on post-operative days one and two
* Presence/Absence of Bowel/Bladder Function

Data to be Collected by Physical Therapist: POD 1, 2, 3, Numerical Rating Scale (NRS) Pain with Ambulation

* Use of Assisted Devices
* Distance walked
* Range of Motion(ROM) (using Goniometer)- active and passive.

Treatment Periods Screening Visit Day 0 - Day of surgery Visit Day 1, 2, 3 (Post-operative days 1, 2, and 3) 6 Week visit in Office

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women aged 30 to 85 years
2. Voluntary, written informed consent given to participate in this clinical investigation

Exclusion Criteria:

1. Pregnant or lactating women
2. Presence of allergies or contraindication to any medications indicated in the study
3. Contraindication to or failure of spinal anesthesia
4. Known drug or alcohol abuse or psychologic disorder that could affect follow-up care or treatment outcomes
5. Patients with a diagnosis of inflammatory arthritis
6. Previous major bone surgery in the operative knee
7. Simultaneous, bilateral TKRs

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F. Dalury, MD, Principal Investigator — Towson Orthpaedic Associates

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients scheduled for Total Knee Replacement (TKR), by the investigator and considered suitable for participation,were recruited for the study from Jan 2010 through June 2011.
Pre-assignment Details: Before assignment to groups all participants were screened for certain exclusion criteria including; pregnant/lactating women, allergies/contraindications to study medications/spinal anesthesia, drug/alcohol abuse, psychologic disorder, diagnosis of inflammatory arthritis, previous major surgery to operative knee, and simultaneous bilateral TKR's.
Groups:
- ROP/EPI/TOR/CLO: Ropivicaine 5mg/ml (49.25 ml) Epinephrine 1 mg/ml (0.5 ml) Toradol 30mg/ml (1 ml) Clonidine 0.1 mg/ml (0.08mg - 0.8 ml)
- REP/EPI/TOR: Ropivicaine 5mg/ml (49.25 ml) Epinephrine 1 mg/ml (0.5 ml) Toradol 30mg/ml (1 ml)
- REP/EPI/CLO: Ropivicaine 5mg/ml (49.25 ml) Epinephrine 1 mg/ml (0.5 ml) Clonidine 0.1 mg/ml (0.08mg - 0.8 ml)
- REP/EPI: Ropivicaine 5mg/ml (49.25 ml) Epinephrine 1 mg/ml (0.5 ml)
Period: Overall Study
Arm/Group | ROP/EPI/TOR/CLO | REP/EPI/TOR | REP/EPI/CLO | REP/EPI
Started | 40 | 40 | 40 | 40
Completed | 38 | 38 | 38 | 36
Not Completed | 2 | 2 | 2 | 4
Not completed — Protocol Violation | 2 | 2 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- ROP/EPI/TOR: Ropivicaine 5mg/ml (49.25 ml) Epinephrine 1 mg/ml (0.5 ml) Toradol 30mg/ml (1 ml)
- ROP/EPI/CLO: Ropivicaine 5mg/ml (49.25 ml) Epinephrine 1 mg/ml (0.5 ml) Clonidine 0.1 mg/ml (0.08mg - 0.8 ml)
- ROP/EPI: Ropivicaine 5mg/ml (49.25 ml) Epinephrine 1 mg/ml (0.5 ml)
- Total: Total of all reporting groups
Arm/Group | ROP/EPI/TOR/CLO | ROP/EPI/TOR | ROP/EPI/CLO | ROP/EPI | Total
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 19 | 16 | 11 | 59
  >=65 years | 27 | 21 | 24 | 29 | 101
Age Continuous [Mean (Standard Deviation); unit: years] | 66.74 (8.07) | 66.29 (8.20) | 68.26 (7.47) | 69.25 (8.67) | 67.64 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 25 | 27 | 98
  Male | 17 | 17 | 15 | 13 | 62
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 40 | 40 | 160

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale (NRS) Pain Scores During Hospitalization.
Description: Patient pain was assessed during hospitalization using the VAS Pain Scale, a numerical rating scale ranging from 0 (no pain) to 10 (severe pain). A lower score represents a better outcome. Pain was assessed preoperatively, 1 hour postoperatively in the post anesthesia unit, and then every 8 hours on the Orthopedic inpatient unit, for a duration of 2 days.
Time Frame: 2 days after surgery
Measure: Mean (Standard Deviation); unit: scores on a scale 0-10
Arm/Group | ROP/EPI/TOR/CLO | ROP/EPI/TOR | ROP/EPI/CLO | ROP/EPI
Number analyzed (Participants) | 38 | 38 | 38 | 36
scores on a scale 0-10
  Vas Pain Scale - 1 Hour Post Op | 1.06 (1.74) | 1.90 (1.04) | 2.67 (3.06) | 1.60 (2.01)
  Vas Pain Scale - 8 Hour Post Op | 1.52 (1.54) | 1.52 (1.56) | 3.93 (2.57) | 2.82 (1.93)
  Vas Pain Scale - 16 Hour Post Op | 1.85 (1.69) | 2.22 (2.36) | 2.75 (2.36) | 2.41 (1.65)
  Vas Pain Scale - 24 Hour Post Op | 2.33 (2.06) | 2.56 (1.76) | 3.63 (2.86) | 2.96 (2.28)
  Vas Pain Scale - 32 Hour Post Op | 2.18 (2.13) | 2.66 (2.13) | 3.62 (2.19) | 3.13 (2.07)
  Vas Pain Scale - 40 Hour Post Op | 2.54 (2.20) | 2.35 (2.31) | 3.28 (2.49) | 2.80 (2.27)
  Vas Pain Scale - 48 Hour Post Op | 2.41 (2.25) | 1.97 (1.72) | 2.56 (2.20) | 2.11 (1.98)
  Vas Pain Scale Preoperatively | 1.93 (2.07) | 2.47 (2.25) | 2.43 (2.40) | 2.13 (2.48)

2. Secondary Outcome: Narcotic Consumption During Hospitalization
Description: A variety of pain medications were used after surgery to keep patients comfortable. Narcotic use was recorded as morphine equivalents. We report the mean narcotic consumption for each group for the day of surgery as well as post operative day 1,2, and 3.
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | ROP/EPI/TOR/CLO | ROP/EPI/TOR | ROP/EPI/CLO | ROP/EPI
Number analyzed (Participants) | 38 | 38 | 38 | 36
mg
  Morphine Equivalent Day of Surgery | 46.92 (22.29) | 43.09 (25.33) | 55.20 (28.00) | 52.50 (27.12)
  Morphine Equivalent Post Operative Day 1 | 46.54 (29.14) | 47.95 (35.89) | 64.61 (41.71) | 51.08 (39.98)
  Morphine Equivalent Post Operative Day 2 | 40.71 (29.67) | 42.69 (37.28) | 50.07 (44.11) | 36.76 (35.28)
  Morphine Equivalent Post Operative Day 3 | 20.45 (19.88) | 18.72 (20.73) | 21.97 (22.38) | 15.54 (21.77)

3. Secondary Outcome: Knee Society Pain Scores at 6 Week Follow-up Appointment
Description: Patients were assessed for pain at their 6 week follow-up appointment using the Knee Society Rating Scale. Using this scale patients are given a pain score ranging from 0 (severe pain) to 50 (No Pain). This is determined as follows: No pain/50 points, Mild or occasional pain/45 points, pain with stairs only/40 points, pain with walking and stairs/30 points, Moderate/occasional pain/ 20 points,continual pain/10 points, severe pain/0 points. We report the mean score for each group. A higher score represents a better outcome.
Time Frame: 6 weeks after surgery
Measure: Mean (Full Range); unit: Scores on a scale 0-50
Arm/Group | ROP/EPI/TOR/CLO | REP/EPI/TOR | REP/EPI/CLO | REP/EPI
Number analyzed (Participants) | 38 | 38 | 38 | 36
Scores on a scale 0-50 | 45 [30 to 50] | 43 [10 to 50] | 45 [10 to 50] | 45 [10 to 50]

ADVERSE EVENTS:
Arm/Group | ROP/EPI/TOR/CLO | ROP/EPI/TOR | ROP/EPI/CLO | ROP/EPI
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes